CLINICAL TRIAL: NCT00426153
Title: Pilot Study Of Long-Acting Octreotide (Octreotide LAR® Depot) In The Treatment Of Patients With Severe Polycystic Liver Disease
Brief Title: Octreotide in Severe Polycystic Liver Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Novartis (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Marie Hogan, MD, PhD, Assistant Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-004128; UL1RR024150 (NIH)
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Polycystic Kidney, Autosomal Dominant; Polycystic Liver Disease; Hepatomegaly; Liver Diseases; Kidney, Polycystic; Abdominal Pain
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic liver disease; Hepatomegaly; Liver Diseases; Polycystic Kidney Diseases; Abdominal Pain | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octreotide (Active Comparator): Participants received Octreotide LAR® Depot injections (up to 40 mg) intramuscularly every 28 days (+/- 5 days) for one year
  Interventions: Drug: Octreotide
- Placebo (Placebo Comparator): Participants received an injection of placebo (sham) medication intramuscularly every 28 days (+/- 5 day) for one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Participants received Octreotide LAR® Depot injections (up to 40 mg)intramuscularly every 28 days (+/- 5 days) for one year
  Other Names: Octreotide LAR® Depot
  Arms: Octreotide
Drug: Placebo — Participants received an injection of placebo (sham) medication intramuscularly every 28 days (+/- 5 day) for one year
  Other Names: Placebo injection
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of Octreotide LAR® on the liver volumes of patients with severe polycystic liver disease who are not candidates or decline surgical treatments such as liver cyst fenestration, liver resection or liver transplantation. A total of 42 patients will be recruited -14 who will receive placebo and 28 the study drug. Preliminary evidence indicates that this drug is safe and non-toxic in other disease states. Treatment with this drug holds promise not only for individuals with liver involvement, but also for many more patients with polycystic kidney disease.

DETAILED DESCRIPTION:
The primary aim of this study is to compare the effect of Octreotide LAR® Depot on the liver volume of patients with severe polycystic liver disease who are not candidates or decline surgical treatments such as liver cyst fenestration, liver resection or liver transplantation compared with placebo. The secondary aims of the study are: (1)Assess the effect of Octreotide LAR® Depot on the total kidney volume and iothalamate clearance in patients with polycystic kidney disease associated with severe polycystic liver disease who are not candidates or decline surgical treatments such as liver cyst fenestration, liver resection or liver transplantation. (2)Evaluate quality of life changes associated with the administration of Octreotide LAR® Depot in these patients. (3)Assess toxicity of Octreotide LAR® Depot in patients with polycystic liver disease (PLD).

Note: Subjects who completed this 1 year randomized trial were offered enrollment into an open-label (all subjects received Octreotide) extension trial for an additional two years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years and older
* Diagnosis of Polycystic Liver Disease (PLD) associated with ADPKD or isolated Autosomal Dominant Polycystic liver Disease (ADPLD)
* Severe PLD defined as a liver volume greater than 4000 mL or symptomatic disease due to mass effects from hepatic cysts
* Not a candidate for or declining surgical intervention

Exclusion Criteria:

* Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception
* Creatinine greater than 3mg/dL or hemodialysis dependent
* Cancer or major systemic disease that could prevent completion of the planned follow-up or interfere with data collection or interpretation
* Uncontrolled diabetes mellitus as defined by blood glucose levels of greater than or equal to 250 mg/dL on 2 or more consecutive daily readings despite antidiabetic therapy
* Neurologic/psychologic conditions preventing appropriate informed consent
* Symptomatic gallstones or biliary sludge
* Variceal bleeding or hepatic encephalopathy within prior 30 days
* Uncontrolled hypertension (Systolic blood pressure greater than 160 mmHg; Diastolic blood pressure greater than 100 mmHg)
* Current, or prior use of somatostatin analogue (octreotide, lanreotide) in past 6 months
* History of significant adverse reaction to a somatostatin analogue

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie C. Hogan, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Hogan MC, Masyuk TV, Page L, Holmes DR 3rd, Li X, Bergstralh EJ, Irazabal MV, Kim B, King BF, Glockner JF, Larusso NF, Torres VE. Somatostatin analog therapy for severe polycystic liver disease: results after 2 years. Nephrol Dial Transplant. 2012 Sep;27(9):3532-9. doi: 10.1093/ndt/gfs152. Epub 2012 Jul 6. PMID 22773240
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Hogan MC, Masyuk T, Bergstralh E, Li B, Kremers WK, Vaughan LE, Ihrke A, Severson AL, Irazabal MV, Glockner J, LaRusso NF, Torres VE. Efficacy of 4 Years of Octreotide Long-Acting Release Therapy in Patients With Severe Polycystic Liver Disease. Mayo Clin Proc. 2015 Aug;90(8):1030-7. doi: 10.1016/j.mayocp.2015.05.011. Epub 2015 Jul 9. PMID 26166166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 participants were enrolled at Mayo Clinic in Rochester, Minnesota from 1/1/2007 to 5/19/2008.
Pre-assignment Details: Following consent a tolerability test dose of 100 micrograms of short-acting octreotide was administered subcutaneously to subjects, followed by 4 hours of observation/vital signs. Randomized intramuscular dosing began the next day.
Groups:
- Octreotide: Participants received Octreotide LAR® Depot injections intramuscularly every 28 days (+/- 5 days) for one year
Period: Overall Study
Arm/Group | Octreotide | Placebo
Started | 28 (Participants were randomized in a 2:1 ratio, Octreotide LAR depot: Placebo) | 14
Completed | 28 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide | Placebo | Total
Number analyzed (Participants) | 28 | 14 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 49.7 (9) | 50.3 (7.3) | 49.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 28 | 14 | 42
Glomerular Filtration Rate [Mean (Standard Deviation); unit: milliliters/minute per 1.73 m^2] — Glomerular Filtration Rate measures how fast the kidneys are filtering. 13 subjects were excluded from the analysis of the kidney data: 4 subjects had renal transplant before enrollment (3 in octreotide and 1 in placebo groups), 8 subjects had a diagnosis of ADPLD (4 in each group), 1 placebo subject has missing kidney data due to incomplete image coverage.
  milliliters/minute per 1.73 m^2 | 70 (27) | 71 (27) | 70 (27)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kilograms/meter^2 | 26.3 (5.77) | 24.4 (2.98) | 25.7 (5.0)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 76.0 (20.2) | 70.9 (10.9) | 74.3 (17.8)
Serum creatinine [Mean (Standard Deviation); unit: milligrams/deciliter] — Creatinine in the serum is a blood test, and is an indicator of kidney function.
  milligrams/deciliter | 1.1 (0.4) | 1.1 (0.5) | 1.1 (0.5)
Fasting plasma glucose [Mean (Standard Deviation); unit: milligrams/deciliter] | 93.4 (11.2) | 93.6 (7.8) | 93.5 (10.1)
Urine Albumin [Mean (Standard Deviation); unit: milligrams/24 hours] — A protein urine test measures the amount of proteins, such as albumin, found in a urine sample. Urine albumin is an indicator of kidney function.
  milligrams/24 hours | 65 (123) | 130 (237) | 87 (171)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Systolic blood pressure is the upper number on a blood pressure reading and measures contraction of the ventricles, or lower chambers of the heart
  millimeters of mercury (mmHg) | 122.1 (13.2) | 120.5 (13.5) | 121.6 (13.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Diastolic blood pressure is the lower number on a blood pressure reading and measures dilation of the ventricles, or lower chambers of the heart.
  millimeters of mercury (mmHg) | 79.8 (8.9) | 79.1 (9.2) | 79.6 (8.9)
Liver volume [Mean (Standard Deviation); unit: milliliters (ml)] — Liver volume was measured by magnetic resonance imaging (MRI) or computed tomography [CT].
  milliliters (ml) | 5907.7 (2915.0) | 5373.9 (3565.4) | 5729.8 (3113.1)
Kidney volume [Mean (Standard Deviation); unit: milliliters (ml)] — Kidney volume was measured by magnetic resonance imaging (MRI) or computed tomography [CT].
  13 subjects were excluded from the analysis of the kidney data: 4 subjects had renal transplant before enrollment (3 in octreotide and 1 in placebo groups), 8 subjects had a diagnosis of ADPLD (4 in each group), 1 placebo subject has missing kidney data due to incomplete image coverage. (Octreotide group n = 21 and placebo group n = 8).
  milliliters (ml) | 1142.9 (826.9) | 803.0 (269.1) | 1049.2 (728.3)
Genotypes and genetic mutations [Number; unit: Participants] — Autosomal dominant polycystic kidney disease (ADPKD) is caused by mutations in one of two genes: PKD1 or PKD2, and is characterized by the development of kidney cysts and other manifestations, of which polycystic live disease (PLD) is most common. Autosomal dominant PLD (ADPLD) also exists as a genetically distinct disease with few or absent kidney cysts. Like ADPKD, ADPLD is genetically heterogeneous, with the 1st two genes identified (PRKCSH & SEC63) accounting for approximately 1/3 to 1/2 of isolated ADPLD cases.
  Participants
    ADPKD genotype with PKD1 gene mutation | 16 | 9 | 25
    ADPKD genotype with PKD2 gene mutation | 5 | 1 | 6
    ADPKD genotype with no genetic mutation detected | 3 | 0 | 3
    ADPLD genotype with PRKCSH gene mutation | 3 | 1 | 4
    ADPLD genotype with SEC63 gene mutation | 0 | 1 | 1
    ADPLD genotype with no genetic mutation detected | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Liver Volume
Description: Percent change from baseline in liver volume, measured in milliliters by Magnetic Resonance Imaging (MRI)or Computed Tomography (CT) scans
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 28 | 14
percent change | -5.0 (6.77) | 0.9 (8.33)
Statistical Analysis 1: Comparison: Octreotide vs Placebo; P values <0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.048, Rank-sum test

2. Secondary Outcome: Percent Change in Renal Volume
Description: Percent change from baseline in renal volume, measured in milliliters by MRI or CT scans
Time Frame: Baseline, 12 months
Population: 13 subjects were excluded from the analysis of the kidney data: 4 subjects had renal transplant before enrollment (3 in octreotide and 1 in placebo groups), 8 subjects had a diagnosis of ADPLD (4 in each group), 1 placebo subject has missing kidney data due to incomplete image coverage.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 21 | 8
percent change | 0.25 (7.53) | 8.61 (10.07)
Statistical Analysis 1: Comparison: Octreotide vs Placebo; Test type: Superiority or Other; p = 0.045, Rank sum — P values < 0.05 were considered statistically significant

3. Secondary Outcome: Percent Change in Glomerular Filtration Rate (GFR)
Description: Percent change from baseline in renal function/GFR, measured by clearance of iothalamate with monitoring of bladder emptying using ultrasound
Time Frame: Baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 21 | 8
percent change | -5.1 (15.46) | -7.2 (13.21)
Statistical Analysis 1: Comparison: Octreotide vs Placebo; Test type: Superiority or Other; p = 0.98, Rank sum — P Values < 0.05 were considered statistically significant

4. Secondary Outcome: Change in Subject Reported Outcomes Using Mean Health Related Quality of Life (HRQoL) Scores
Description: Scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36), version 2. Subjects completed the SF-36 which consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 24 | 12
units on a scale
  Physical functioning at baseline | 74.8 (21.96) | 80.4 (23.73)
  Physical functioning at 12 months | 77.0 (21.32) | 82.1 (18.58)
  Physical role at baseline | 59.8 (42.13) | 76.8 (39.79)
  Physical role at 12 months | 74.1 (35.00) | 75.0 (41.60)
  Bodily Pain at baseline | 67.8 (15.29) | 65.5 (24.25)
  Bodily pain at 12 months | 75.7 (19.02) | 68.7 (25.51)
  General health at baseline | 55.9 (21.29) | 58.0 (23.63)
  General health at 12 months | 53.5 (17.32) | 63.4 (23.96)
  Vitality at baseline | 49.6 (21.81) | 53.9 (25.96)
  Vitality at 12 months | 54.4 (24.23) | 54.6 (27.91)
  Social functioning at baseline | 79.0 (19.56) | 75.0 (27.30)
  Social functioning at 12 months | 82.9 (19.35) | 81.3 (21.79)
  Emotional role at baseline | 82.1 (32.05) | 73.8 (37.39)
  Emotional role at 12 month | 91.4 (23.74) | 81.0 (38.60)
  Mental health at baseline | 76.0 (14.12) | 75.4 (18.75)
  Mental health at 12 months | 76.9 (16.54) | 80.7 (18.76)
  Standardized physical component at baseline | 42.6 (9.73) | 46.0 (10.16)
  Standardized physical component at 12 months | 44.7 (10.00) | 46.1 (9.51)
  Standardized mental component at baseline | 50.8 (7.74) | 48.4 (10.96)
  Standardized mental component at 12 month | 52.2 (8.03) | 51.3 (11.15)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Octreotide | Placebo
Serious Adverse Events (participants affected / at risk) | 3/28 | 0/14
Other Adverse Events (participants affected / at risk) | 21/28 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=28) | Placebo (N=14)
Abdominal hernia, incarcerated (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hernia surgically repaired
Bacteremia (Renal and urinary disorders) | 1 (1) | 0 (0) — Bacteremia associated with nephrolithiasis
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — UTI, abdominal pain and fever responded to antibiotic therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=28) | Placebo (N=14)
Alopecia, moderate (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea, Grade 1 (Gastrointestinal disorders) | 17 (17) | 4 (4)
Injection site granuloma (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Injection site pain (Skin and subcutaneous tissue disorders) | 21 (21) | 3 (3)
Steatorrhea & weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject withdrew from study due to steatorrhea & weight loss
abdominal cramping, bloating and gas (Gastrointestinal disorders) | 14 (14) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No